CLINICAL TRIAL: NCT00900055
Title: Dysregulation of Hematopoiesis in Fanconi Anemia
Brief Title: Research Study in Healthy Volunteers of Patients With Fanconi Anemia, Myeloproliferative Disorders, or Myeloma
Status: Completed | Type: Observational
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Laura Newell, Assistant Professor, OHSU Knight Cancer Institute
Other Study IDs: IRB00000823; P01HL048546 (NIH); OHSU-HEM-98030-L
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Chronic Myeloproliferative Disorders; Fanconi Anemia; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic/Myeloproliferative Neoplasms
Keywords: Fanconi anemia; multiple myeloma and other plasma cell neoplasms; chronic myeloproliferative disorders; myelodysplastic/myeloproliferative neoplasms
MeSH Terms: conditions — Myeloproliferative Disorders; Fanconi Anemia; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic-Myeloproliferative Diseases | interventions — Microarray Analysis; Electrophoresis, Polyacrylamide Gel; Polymerase Chain Reaction; Reverse Transcriptase Polymerase Chain Reaction; Blotting, Western; Chromatography; Chromatography, High Pressure Liquid; Immunoenzyme Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Genetic: microarray analysis
Genetic: polyacrylamide gel electrophoresis
Genetic: polymerase chain reaction
Genetic: protein expression analysis
Genetic: reverse transcriptase-polymerase chain reaction
Genetic: western blotting
Other: chromatography
Other: high performance liquid chromatography
Other: immunoenzyme technique

SUMMARY:
RATIONALE: Analyzing tissue and blood samples from healthy volunteers or patients with Fanconi anemia, myelodysplasia, myeloproliferative disorders, or myeloma in the laboratory may help doctors learn more about the causes of blood cancers.

PURPOSE: The purpose of this study is to analyze in the laboratory blood and bone marrow cells from healthy volunteers or patients with Fanconi anemia, myeloproliferative disorders, or myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Identify the specific molecular function of the Fanconi anemia (FA) complementing gene products in hematopoietic progenitor cells from patients and normal volunteers.
* Identify functional defects in hematopoietic stromal cells, including macrophages, from patients with FA, and selected blood cancers as well as normal volunteers.

OUTLINE: Peripheral blood mononuclear leukocytes, skin fibroblasts, and marrow fibroblasts are collected for loss-of-function and gain-of-function analysis related to the Fanconi anemia complementing gene.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * Diagnosis of one of the following:

    * Fanconi's anemia requiring bone marrow biopsy as part of standard care (adults and children)
    * Myeloproliferative disorder or myeloma (adults)
  * Healthy volunteer, meeting 1 of the following criteria:

    * Over 18 years of age
    * Bone marrow transplant donor (children)

PATIENT CHARACTERISTICS:

* Hemoglobin > 13 g/dL
* White blood cells (WBC) > 4,000/mm³
* Platelet count > 150,000/mm³
* No clinical signs or symptoms of acute or subacute infections (viral, bacterial, or fungal)
* No known blood abnormality (healthy volunteers)
* No allergies to lidocaine or xylocaine

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 1 Year to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The Center for Hematologic Malignancies, the Knight Cancer Institute at OHSU, and the Bone Marrow Failure clinic at Doernbecher Children's Hospital at OHSU will be centers for recruitment.
Sampling Method: Probability Sample
Enrollment: 213 (Actual)
Dates: Start 1975-06; Primary Completion 2016-08-23 (Actual); Study Completion 2016-08-23 (Actual)

PRIMARY OUTCOMES:
Loss of function analyses | Duration of the study
Proteins binding to Fanconi anemia, complementation group C (FACC) gene-product by affinity chromatography of nuclear and whole cell lysates of normal cells | Duration of the study
Screening of proteins binding to FACC gene-product using monoclonal antibodies specific to signal transduction and cell cycle proteins | Duration of the study
Microsequencing of unique proteins | Duration of the study
Location of specific downstream block point imposed by antisense molecules using antibodies specific to signal transduction, cell cycle, or repair proteins for the FACC protein | Duration of the study
Affirmation that the block points identified are recapitulated in progenitor cells from peripheral blood | Duration of the study
Identification of functional defects in Fanconi anemia hematopoietic stromal cells | Duration of the study

CONTACTS AND LOCATIONS:
Overall Officials: Laura Newell, MD, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- Knight Cancer Institute at Oregon Health and Science University, Portland, Oregon, United States